CLINICAL TRIAL: NCT06664229
Title: Development of the Flexible and Printed Electronic Device for Dementia and Fall Prevention of Older Adults
Brief Title: Development of Pressure Sensor Based Dementia and Fall Prevention Program for Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunmi Song (Other)
Responsible Party: Sponsor-Investigator, Sunmi Song, Research Professor, Korea University
Organization: Korea University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Q2317781
Record Dates: First submitted 2024-03-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Dementia, Mild; Accidental Falls; Mild Cognitive Impairment
Keywords: Fall prevention; Dementia prevention; Mild cognitive impairment; Exercise game; Cognitive training game; Community based intervention; Older adults
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Cognitive Dysfunction | interventions — Accidental Falls

STUDY DESIGN:
Intervention Model Description: We will conduct a single-blind randomized control trial design for the main study. The pilot study will have the intervention group only without the control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be research assistants who do not know the group assignment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Older adults who participated in a group exercise program using the developed mat and software three times per week for six weeks (18 sessions) for a pilot study and twelve weeks (36 sessions) for a main study took part in the pre-post tests. The frequency and duration can be adjusted to twice per week for nine weeks (18 sessions) for a pilot study or twice per week for sixteen weeks (32 sessions) for a main study to accommodate the availability of participants and the spaces in the community center.
  Interventions: Behavioral: Fall and dementia prevention exercise
- Control group (No Intervention): Older adults who participated only in the pre-post tests without receiving any intervention.

INTERVENTIONS:
Behavioral: Fall and dementia prevention exercise — The fall and dementia prevention exercise is designed as a combination of balancing and cognitive exercise and games that is conducted as a group activity. The session will be provided three times per week for six weeks for a pilot test and three times per week for 12 weeks for a main comparison study.
  The fall prevention exercise involves the pressure mat based balancing exercise such as side stepping, heel or toe standing, and quarter squat. The safety bar will be placed around the mat, so that older adults with instability can hold while they follow the movements.
  The cognitive exercise will concise of multiple types of cognitive tasks to train memory, numeric processing, spatial perception, and logical thinking. For example, memory task such as memorizing the series of positions on the screen and use the mat to point the positions in the right order.
  At the end, older adults play games in which they use balancing movements and cognitive tasks to gain scores for their team.
  Arms: Intervention group

SUMMARY:
The goal of this intervention program is to test the effectiveness of pressure sensor based dementia and fall prevention program for improving cognitive and physical functions of community dwelling older adults. The main purposes of this study are:

1. Develop a pressure sensor based exercise mat and linked software programs to be used for group training sessions for cognitive and balance training of older adults at a community senior center.
2. Evaluate efficacy of the program to improve cognitive and physical functions of older adults via a pilot study and a main study with randomized control trial design.

Older adults will be asked to participate in a group training session that was lead by a fitness coach using a pressure sensor mat, a standing monitor, and a linked software programs. They will be asked to stand on the mat, which is set in front of a monitor to show positions of the mat where they place their foots. The monitor screen will guide them to conduct either a balancing exercise for fall prevention or a cognitive exercise such as memory game or quiz game for dementia prevention.

Researchers will compare age and gender matched control group in a main study to see if cognitive and balancing functions of intervention group is better than the control group by conducting pre and post surveys and physical examinations. A pilot study will examine pre-post changes in the intervention group without the control group.

DETAILED DESCRIPTION:
A. Developed group exercise devices

○ The study will test the flexible, stretchable film-type pressure sensor embedded balance mat and a monitor that will present a sequence of fitness programs and cognitive tasks.

* A 65cm wide balance mat embedded with pressure sensors will be utilized for balance trainings and responding to cognitive tasks.
* The devices are consisted of hardware and software based on a thin, flexible pressure sensor (includes additional safety aids such as safety bars and surrounding cushion mats).
* The thin pressure sensor allows for a lightweight, portable mat.

B. Pilot Test

* The pilot test will be conducted with a single intervention group who participated in the group exercises using the developed devices that are led by a trainer.
* Pre- and post-assessment: Two measurements will be taken before and after the intervention, evaluating balance, physical fitness, cognition, and quality of life.
* User-centered interviews: One interview will be conducted after the intervention to gather participants' opinions on the exercise program and to determine the direction of future studies. The interview will use the Metaplan method, which was verified as an effective approach for developing assistive systems for older users in a previous study (Thoma-Lürken et al., 2018). The interview will be conducted with four participants from the pilot test, and the interview session will last 60 to 90 minutes, considering participants' needs for breaks. For effective data collection and analysis, the entire interview process will be recorded with participants' prior consent.

C. The main test

* The main test will be conducted with single-blind, randomized controlled trial (RCT) design. The intervention group will participate in the group exercises using the developed devices that are led by a trainer.

  * Random assignment: Block randomization (block size 4) will be applied to randomly assign participants to the intervention group or the control group.
  * Single-blind (blinding of the evaluator): The evaluator will not be informed of the participants' group allocation during assessments.
* Pre-, mid-, and post-assessment: Measurements will be taken three times-before the intervention, after 8 weeks of exercise, and after 16 weeks of exercise-assessing balance, physical fitness, cognition, depression, sleep, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Older adults in the community who are 65 years old or older.

Exclusion Criteria:

* Older adults who cannot walk independently with assisting devices or use wheelchair.
* Older adults who are diagnosed with dementia, or other neurological/mental disorders that may limit their cognitive ability to participate in the study.
* Older adults who cannot speak or read Korean.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Berg Balance test | The Berg balance test will be conducted at baseline (one week before the first session), mid-term survey (6th week of 12 week program or 8th week of 16 week program), and within one week following the last session of the intervention (13th or 17th week).
  The Berg Balance test (Lusardi, 2004) ranges from 0 to 56 with lower score indicating the more risk of losing one's balance.
The Mini-Mental State Exam Korean Version (MMSE-K) | The system usability test will be conducted at baseline and within one week following the last session of the intervention.
  The Mini-Mental State Exam Korean version (MMSE-K) ranges from 0-30 with higher score indicating better cognitive function.
The Morse Fall Risk Scale | The system usability test will be conducted at baseline and within one week following the last session of the intervention.
  The Morse Fall Risk Scale ranges 0-125 with higher score indicating higher risk of fall.
Montreal Cognitive Assessment (MoCA) | MoCA will be conducted at baseline and within one week following the last session of the intervention.
  MoCA test will be conducted to examine changes in cognitive functioning before and after the intervention program.
Grip test | The grip test will be conducted at baseline, and at the mid-term assessment, and within one week following the last session of the intervention.
  A test that measures left and right grip strength (kg). The larger the test score, the stronger the grip strength.
The 30 second sit-stand test | The 30 second sit-stand test will be conducted at baseline, mid-term survey, and within one week following the last session of the intervention.
  The 30 second sit-stand test measures the number of completed chair stands in 30 seconds. The larger number of completed chair stands, the better physical fitness of a participant.
The 2 minute step in place test | The 2 minute step in place test will be conducted at baseline, mid-term survey, and within one week following the last session of the intervention.
  The 2 minute step in place test (number): A test that measures the total number of times the right knee reaches the tape level in two minutes. The more number of reaches, the better fitness scores the participant has.
The sit and reach test (cm) | The sit and reach test will be conducted at baseline, mid-term survey, and within one week following the last session of the intervention.
  The sit and reach test (cm) measures the distance reached by the hand. The participant sits on the floor with legs stretched out straight ahead, with the soles of the feet flat against the box. Both knees should be locked and pressed flat to the floor. Reach forward with a slow and steady movement as far as possible, and hold that position for three seconds while the distance is recorded. The larger scores indicate the better fitness of the participant.
The 3 m sit-walk and return test | The 3 m sit-walk and return test will be conducted at baseline, mid-term survey, and within one week following the last session of the intervention.
  The 3 m sit-walk and return test measures the time (seconds) from sitting on a chair to standing, walking to a 3 m target, and then returning to the chair and sitting down. The shorter test score indicates better fitness of a participant.
The figure of 8 walk test | The figure of 8 walk test will be conducted at baseline, mid-term survey, and within one week following the last session of the intervention.
  The figure of 8 walk test measures the time (seconds) to walk a figure-of-eight around 2 cones placed 2.4 m apart twice. The smaller score indicates the better walking ability of a participant.

SECONDARY OUTCOMES:
Geriatic depression | Geriatric depression scale will be conducted at baseline and within one week following the last session of the intervention.
  Geriatric depression scale score ranges from 0-15 with higher scores indicating more severe depressive symptoms.
Pain related functional limitations | The WOMAC will be conducted at baseline and within one week following the last session of the intervention.
  The brief version of the Western Ontario and McMaster Universities Osteoarthritis Index, which measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68), with higher scores indicating worse pain and functional limitations in one's daily living.
The Pittsburgh Sleep Quality Index (PSQI) | The PSQI will be conducted at baseline, mid-term survey, and within one week following the last session of the intervention.
  The brief version of the Pittsburgh Sleep Quality Index ranges from 0 to 15 with higher score indicating more sleep problems.
WHO quality of life bref | The system usability test will be conducted at baseline and within one week following the last session of the intervention.
  WHO quality of life bref assesses physical, psychological, social, environmental health, which ranges 7-35, 6-30, 3-15, 8-40, respectively, higher score indicating better physical, psychological, social, environmental health status.

OTHER OUTCOMES:
System Usability Test | The system usability test will be conducted at baseline, mid-term survey, and within one week following the last session of the intervention.
  System usability test will be conducted to examine changes in the levels of usability for the digital devices that were developed for the intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Junesun Kim, PT/PhD, Principal Investigator — Korea University
Locations (1):
- Korea University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The IRB approval of this study do not allow sharing data from this study with other researchers.